CLINICAL TRIAL: NCT04068935
Title: Buddy Taping Compared to Splint Immobilizations for Reduced Paediatric Finger Fractures
Brief Title: Buddy Taping Compared to Splint Immobilization for Displaced Paediatric Finger Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Buddy taping 2019
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Fracture Finger

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buddy taping (Experimental): Buddy taping of the fractured finger to ist neighbouring uninjured finger.
  Interventions: Procedure: fracture immobilization after reduction of displaced finger fractures
- splint immobilization (Active Comparator): A forearm-based palmar Hand Splint in an intrinsic plus Position, enclosing all fingers without the thumb.
  Interventions: Procedure: fracture immobilization after reduction of displaced finger fractures

INTERVENTIONS:
Procedure: fracture immobilization after reduction of displaced finger fractures — After closed reduction of a displaced finger fracture, fracture immobilization with either Buddy taping or Splint immobilization

SUMMARY:
Fracture immobilization with Buddy taping is not inferior to Splint immobilization for non-displaced extra-articular paediatric finger fractures. However, whether the same applies for reduced finger fractures is unclear.

DETAILED DESCRIPTION:
Displaced fractures will be reduced in the paediatric ED by Emergency physicians. After fracture reduction, fracture immobilization will either be done with a Splint immobilization or a fingertaping. After 4 and 21 days, clinical and radiographic controls will take place at the Hand surgery outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* extraarticular displaced finger fractures of the proximal or middle phalanges

Exclusion Criteria:

* fractures of the thumb
* fractures that are open, instable, pathologic or multifragmented
* multiple fractures of the Hand
* phalangeal neck fractures
* presentation later than 5 days after the injury

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
secondary fracture displacement | 5 and 21 days after fracture reduction
  X-ray controls

SECONDARY OUTCOMES:
Patient comfort | 5 and 21 days after fracture reduction
  visual analog scale (VAS): Smiley scale with a range from 1 to 10, 10 being the highest score possible, indicating that the Patient comfort was very high.
Need for analgesic medication | 5 and 21 days after fracture reduction
  interview with Patient and parents
total range of Motion | 6 month after fracture reduction
  measurement

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Seiler, MD, Principal Investigator — University Children's Hospital, Zurich
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No